CLINICAL TRIAL: NCT03109353
Title: Modification of Extracorporeal Photopheresis Technology With 5-aminolevulinic Acid in Patients With Cutaneous T-cell Lymphoma or Chronic Graft-versus-host Disease - A Proof-of-concept Study
Brief Title: Modification of Extracorporeal Photopheresis in Cutaneous T-cell Lymphoma or Chronic Graft-versus-host Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other); Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-000872-78; 2016-000872-78 (EudraCT Number)
Record Dates: First submitted 2017-04-06; First posted 2017-04-12 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Cutaneous T-Cell Lymphoma, Unspecified; Chronic Graft Versus Host Disease in Skin
Keywords: Photopheresis; 5-aminolevulinic acid; Extracorporeal Circulation
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous | interventions — Eosinophil Cationic Protein; Aminolevulinic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ALA-ECP (Experimental): Extracorporeal photopheresis (ECP) with 5-aminolevulinic acid replacing psoralen
  Interventions: Drug: ECP with 5-aminolevulinic acid

INTERVENTIONS:
Drug: ECP with 5-aminolevulinic acid — extracorporeal photopheresis (ALA-ECP) using 5-aminolevulinic acid instead of psoralen (8-MOP) in a maximum of 10 treatment cycles
  Other Names: 5-ALA

SUMMARY:
Extracorporeal photopheresis (ECP), is commonly used for the treatment of cutaneous T-cell lymphoma (CTCL) and chronic graft-versus-host disease. ECP (cGVHD) is an immune modulating treatment. White blood cells from the patient are standardized activated by a photosensitizer psoralen (8-MOP) and irradiated with visible ultraviolet light (UV-A). The purpose is to induce programmed cell death (apoptosis). Disadvantage of current treatment is that 8-MOP targets both diseased and normal cells with no selectivity.

The purpose of this study is to improve the current ECP technology using aminolevulinic acid (ALA) and UV light. ECP will be carried out in conventional manner except that 8-MOP will be replaced with ALA. Systemic ALA / UV light is already approved and used in the detection and treatment of disease in humans. The primary objective is to assess its safety and tolerability after single and multiple treatment in patients with CTCL or cGvHD.

DETAILED DESCRIPTION:
The main advantages of using ALA for ECP are (1) highly effective and selective apoptotic destruction of transformed/activated hyper-proliferative T-cells through an endogenously selective production of the potent photosensitiser, protoporphyrin IX (PpIX) from ALA via heme biosynthetic pathway; (2) ALA/PpIX only targets membranous structures outside of the cell nucleus thus causing no risk of carcinogenesis and (3) induces systemic anti-tumour immunity.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* cutaneous T-cell lymphoma (CTCL) (Mycosis fungoides and Sézary syndrome)
* considered to respond inadequately to 8-MOP-ECP therapy. Inadequate response is defined as:

  1. progressive disease: disease progression from baseline in skin score, blood or lymph nodes after 3-6 months or
  2. stable disease: No- response after 3-6 months or
  3. minimal response < 50% (from baseline) reduction of skin scores and/or CD4/CD8 ratio or a loss of peripheral blood clone after 3-6 months.
* (or) chronic graft-versus-host disease (cGvHD) and considered to respond inadequately to 8-MOP-ECP therapy. Chronic GvHD is defined as

  1. presence of at least 1 clinical sign of cGvHD or
  2. at least one distinct manifestation confirmed by pertinent biopsy or other relevant tests.
  3. steroid dependence, intolerance or steroid refractoriness considered to respond inadequately to 8-MOP-ECP therapy with at least monthly intervals.

Inadequate response is defined as:

1. progression of cutaneous cGvHD defined as >25% worsening from baseline as measured by the percent change in the total skin score or
2. after 3 months had an inadequate response of cutaneous cGvHD as defined by <15% improvement in the total skin score compared with baseline, or a ≤25% reduction in corticosteroid dose.

Exclusion Criteria:

* Photosensitive comorbidities, porphyria or known hypersensitivity to 5-aminolevulinic acid or porphyrins
* Aphakia
* Pregnancy or breast feeding. (A negative urine pregnancy test must be demonstrated in female patients of child-bearing potential at the Screening Visit)
* Ongoing cardiac and pulmonary diseases or ASAT, ALAT, Bilirubin or INR value ≥ 3x upper limit of normal or clinically significant ECG findings
* Polyneuropathy
* Uncontrolled infection or fever
* History of heparin-induced thrombocytopenia, absolute neutrophil count <1x10-9 L-, platelet count <20x10-9 L-1
* Body weight below 40 kg
* Investigator considers subject unlikely to comply with study procedures, restrictions and requirements.
* History of any clinically significant disease or disorder which in the opinion of the investigator, may either put the patient at risk because of participation in the study, or influence the result or the patient's ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Treatment safety: Monitored through recordings of ECG, vital signs and safety laboratory measurements including haematology, clinical chemistry and urinalysis. | up to 1 year
  Monitored through recordings of ECG, vital signs and safety laboratory measurements including haematology, clinical chemistry and urinalysis.

SECONDARY OUTCOMES:
Main efficacy for CTCL | up to 1 year
  Response of skin disease and reduction in immunosuppression. Response will be evaluated with study baseline as reference as: complete response, partial response, minimal response, stable disease, progressive disease or maximal response based on set definitions.
Main efficacy for cGvHD | up to 1 year
  Response of skin disease and reduction in immunosuppression. Response will be evaluated with study baseline as reference as: complete response, partial response, minimal response, stable disease, progressive disease or maximal response based on set definitions.

CONTACTS AND LOCATIONS:
Overall Officials: Vigleik Jessen, md, Study Director — St Olavs Hospital, Trondheim Unversity Hospital; Torstein Baade Rø, md phd, Study Director — Norwegian University of Science and Technology
Locations (1):
- St Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided